CLINICAL TRIAL: NCT03745794
Title: Randomized Controlled Trial of Repeat vs. Single Quadratus Lumborum Block to Reduce Opioid Prescriptions After Open Pancreatectomy ("RESQU-BLOCK" Trial)
Brief Title: Repeat Quadratus Lumborum Block to Reduce Opioid Need in Patients After Pancreatic Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-0519; NCI-2018-02182 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0519 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-11-14; First posted 2018-11-19 (Actual); Results first posted 2023-02-13 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (QL block, standard of care) (Active Comparator): Patients undergo QL block before surgery and receive standard of care multimodal pain control after surgery.
  Interventions: Other: Best Practice; Drug: Quadratus Lumborum Block; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (second QL block) (Experimental): Patients undergo QL block before surgery and receive multimodal pain control. Patients then undergo a second QL block on day 4 after surgery and continue to receive standard of care.
  Interventions: Other: Best Practice; Drug: Quadratus Lumborum Block; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Given standard of care
  Other Names: standard of care; standard therapy
Drug: Quadratus Lumborum Block — Undergo QL block
  Other Names: QL Block
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how an additional anesthetic nerve block, called a quadratus lumborum block, works to reduce the need for opioids in patients after pancreatic surgery. Giving an additional regional anesthetic after surgery may hasten the weaning process, reduce the need for opioid medications upon discharge, and reduce the risk of opioid dependence.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To use a phase II randomized controlled trial to compare the intervention of a second regional anesthetic block (quadratus lumborum [QL] block) versus usual care (single intraoperative QL block) to increase the proportion of opioid-free pancreatic cancer survivors at discharge after potentially curative surgery.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients undergo QL block before surgery and receive standard of care multimodal pain control after surgery.

ARM 2: Patients undergo QL block before surgery and receive multimodal pain control. Patients then undergo a second QL block on day 4 after surgery and continue to receive standard of care.

After completion of study treatment, patients are followed up at 1 month, 3 months, 6 months, and 1 year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective open pancreatic resection for potentially curative intent (pancreaticoduodenectomy or distal pancreatectomy) who would otherwise be treated with QL block + IV-PCA converted to oral pain meds (non-narcotic bundle + opioid pain pill).

Exclusion Criteria:

* Patients with current or past substance (drug or alcohol) abuse disorder.
* Laparoscopic or minimally invasive surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Wei D Tzeng, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 30 participants were excluded from the study before assignment to arms due to aborted surgery, discharged before 4 days after surgery or opioids free at 3rd day after surgery.
Groups:
- Arm 1, Control Arm (Usual Care): Patients undergo QL block before surgery and receive standard of care multimodal pain control after surgery.
- Arm 2, Experimental Arm (2nd QL-Block): Patients undergo QL block before surgery and receive multimodal pain control. Patients then undergo a second QL block on day 4 after surgery and continue to receive standard of care.
Period: Overall Study
Arm/Group | Arm 1, Control Arm (Usual Care) | Arm 2, Experimental Arm (2nd QL-Block)
Started | 52 | 54
Completed | 52 | 53
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1, Control Arm (Usual Care) | Arm 2, Experimental Arm (2nd QL-Block) | Total
Number analyzed (Participants) | 52 | 53 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 19 | 46
  >=65 years | 25 | 34 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (12.5) | 65 (11.2) | 64 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 47
  Male | 28 | 30 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 8
  Not Hispanic or Latino | 44 | 49 | 93
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 46 | 48 | 94
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 52 | 53 | 105

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Discharged Opioid-Free
Description: Performed Chi-squared test to compare the proportion of patients who were opioid-free on the discharge date between the two arms
Time Frame: 90 days from surgery
Population: one participant inevaluable for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1, Control Arm (Usual Care) | Arm 2, Experimental Arm (2nd QL-Block)
Number analyzed (Participants) | 52 | 53
Participants | 19 | 27
Statistical Analysis 1: Comparison: Arm 1, Control Arm (Usual Care) vs Arm 2, Experimental Arm (2nd QL-Block); Test type: Other; p = 0.17, Chi-squared

2. Secondary Outcome: Total Inpatient Oral Morphine Equivalents (OME)
Description: Two sample t-test or Wilcoxon rank-sum test will be used.
Time Frame: Up to 1 year
Reporting Status: Not Posted, anticipated posting 2026-07

3. Secondary Outcome: Hospital Cost
Description: Two sample t-test.
Time Frame: Up to 1 year
Reporting Status: Not Posted, anticipated posting 2026-07

4. Secondary Outcome: Quality of Life Score Assessed by MD Anderson Symptom Inventory-Gastrointestinal (MDASI-GI)
Description: Two sample t-test or Wilcoxon rank-sum test will be used.
Time Frame: Up to 1 year
Reporting Status: Not Posted, anticipated posting 2026-07

5. Secondary Outcome: Pain Prescription Dosage/Size
Description: Two sample t-test or Wilcoxon rank-sum test will be used.
Time Frame: through study completion, an average of 1 year
Reporting Status: Not Posted, anticipated posting 2026-07

6. Secondary Outcome: Percentage of Patients With Initial Discharge Prescription Dosage/Size Total OME < 200 mg
Description: Two sample t-test or Wilcoxon rank-sum test will be used.
Time Frame: Up to 1 year
Reporting Status: Not Posted, anticipated posting 2026-07

7. Secondary Outcome: Percentage of Patients Using Opioids
Description: Two sample t-test or Wilcoxon rank-sum test will be used.
Time Frame: At 30 days after surgery
Reporting Status: Not Posted, anticipated posting 2026-07

8. Secondary Outcome: MDASI-GI in Clinic Visits
Description: Two sample t-test or Wilcoxon rank-sum test will be used.
Time Frame: Up to 1 year
Reporting Status: Not Posted, anticipated posting 2026-07

9. Secondary Outcome: Percentage of Patients Using Opioids
Description: Two sample t-test or Wilcoxon rank-sum test will be used.
Time Frame: At 90 days after surgery
Reporting Status: Not Posted, anticipated posting 2026-07

10. Secondary Outcome: Total OME for First 30 Days and First 90 Days (Inpatient + Outpatient)
Description: Two sample t-test or Wilcoxon rank-sum test will be used.
Time Frame: At 30 and 90 days
Reporting Status: Not Posted, anticipated posting 2026-07

11. Secondary Outcome: Patients and Family Free of Opioid Use
Description: Two sample t-test or Wilcoxon rank-sum test will be used.
Time Frame: At 6 months and 1 year
Reporting Status: Not Posted, anticipated posting 2026-07

ADVERSE EVENTS:
Time Frame: 90 days from surgery
Description: All surgical complications for 90 days after the surgery were recorded. They were all unrelated to the QL-Block. The MDASI questionnaire survey were collected from 3/1/2019 to 11/29/2021. All deaths were unrelated to the QL-Block.
  In Arm 2, 53 participants were recorded as 1 of the 54 participants dropped out. We were unable to officially track the 90 day outcomes for that participant.
Arm/Group | Arm 1, Control Arm (Usual Care) | Arm 2, Experimental Arm (2nd QL-Block)
All-Cause Mortality (participants affected / at risk) | 3/52 | 3/54
Serious Adverse Events (participants affected / at risk) | 10/52 | 10/54
Other Adverse Events (participants affected / at risk) | 39/52 | 31/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1, Control Arm (Usual Care) (N=52) | Arm 2, Experimental Arm (2nd QL-Block) (N=54)
Delayed Gastric Emptying (Gastrointestinal disorders) | 0 | 1
Pancreatic leak (Gastrointestinal disorders) | 4 | 2
BJ leak (Gastrointestinal disorders) | 1 | 0
Chyle leak (Gastrointestinal disorders) | 0 | 2
GI Other (Gastrointestinal disorders) | 3 | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hemorrhage (Blood and lymphatic system disorders) | 0 | 1
Hematologic_ other (Blood and lymphatic system disorders) | 1 | 0
Abscess (Infections and infestations) | 1 | 2
Sterile collection (Infections and infestations) | 1 | 0
Line infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 0
Infectious Other (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1, Control Arm (Usual Care) (N=52) | Arm 2, Experimental Arm (2nd QL-Block) (N=54)
Delayed Gastric Emptying (Gastrointestinal disorders) | 8 | 7
Pancreatic leak (Gastrointestinal disorders) | 8 | 7
Chyle leak (Gastrointestinal disorders) | 2 | 4
GI Other (Gastrointestinal disorders) | 9 | 3
Arrythmia (Cardiac disorders) | 2 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hemorrhage (Blood and lymphatic system disorders) | 1 | 0
Post-op transfusion (Blood and lymphatic system disorders) | 4 | 5
Hematologic_ other (Blood and lymphatic system disorders) | 2 | 2
Acute Renal Failure (Renal and urinary disorders) | 1 | 0
Renal other (Renal and urinary disorders) | 3 | 3
Abscess (Infections and infestations) | 0 | 1
Cholangitis (Infections and infestations) | 3 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 2
Wound infection (Infections and infestations) | 7 | 2
Colitis (Infections and infestations) | 1 | 0
Infectious Other (Infections and infestations) | 6 | 1
Neurologic_Other (Nervous system disorders) | 1 | 2
Metabolic Other (Metabolism and nutrition disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT03745794/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/94/NCT03745794/ICF_001.pdf